CLINICAL TRIAL: NCT05810675
Title: Parent-mediated and Telehealth Intervention for Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202207134RINB
Record Dates: First submitted 2023-03-20; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder, telehealth, holistic health care
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The intervention group (the telehealth group) will also receive a 16-week telehealth intervention with guidance, digital learning platform, teaching parents to learn intervention skills to improve children's attention and play ability, social communication, cognition, perceptual movement, and improve parents' management of children's behavior problems.
  The comparison group (telephone group) will receive 16-weeks of care and child development counseling through phone calls.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded for the group of participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Early Intervention Program (TEIP) group (Experimental): The TEIP group will also receive a 16-week telehealth intervention with guidance, digital learning platform, teaching parents to learn intervention skills to improve children's attention and play ability, social communication, cognition, perceptual movement, and improve parents' management of children's behavior problems.
  Interventions: Behavioral: Telehealth Early Intervention Program (TEIP)
- Telephone group (No Intervention): The telephone group will receive 16-weeks of care and child development counseling through phone calls.

INTERVENTIONS:
Behavioral: Telehealth Early Intervention Program (TEIP) — The Telehealth Early Intervention Program (TEIP) that will be carried out by parents at home when interact with their children; and to train parents in delivering developmental and behavioral techniques to their children. The participating families will be randomized in parallel to treatment and comparison groups for teaching the knowledge and techniques: (1) Treatment group: providing the training of TEIP for parents via telehealth modalities as they learn critical skills with their child with the goal of increasing multidimensional child developments. Intervention provider will provide the training for parent-child dyad interaction to work with parents to implement these strategies at home environment.
  Other Names: TEIP
  Arms: Telehealth Early Intervention Program (TEIP) group

SUMMARY:
This study has two purposes:

Aim 1: To develop a Telehealth Early Intervention Program (TEIP) for children with ASD that will be carried out by parents at home when interact with their children; and to train parents in delivering developmental and behavioral techniques to their children. The participating families will be randomized in parallel to treatment and comparison groups for teaching the knowledge and techniques: (1) Treatment group: providing the training of TEIP for parents via telehealth modalities as they learn critical skills with their child with the goal of increasing multidimensional child developments. Intervention provider will provide the training for parent-child dyad interaction to work with parents to implement these strategies at home environment; and (2) Comparison group: provide general care consultation of child development for parents.

Aim 2: To evaluate this program's effectiveness by measuring changes in a child's developments and behaviors. Investigator will evaluate child outcomes on the symptoms of ASD and multidimensional developmental functioning. Furthermore, investigator will measure the changes in the parent's knowledge and behaviors of parent-child interaction. Moreover, investigator will determine if parental participation in the intervention is associated with an improvement in parenting competences and decreased levels of stress.

DETAILED DESCRIPTION:
In recent years, due to the rapid increase in the prevalence of autism spectrum disorder (ASD), early detection of these children is helpful for early diagnosis and intervention and better prognosis. Recent research supports the intervention in the daily life of children with autism in a naturalized way. Parents learn intervention skills and implement them in their lives, providing positive effects on children with autism. This type of intervention is called parent-mediated intervention. Pivot Response Training (PRT) is a home-based parent-child intervention model that uses "Applied Behavior Analysis" to integrate into children's daily life situations and teach children to respond appropriately to the many learning opportunities and social interactions in natural situations, reducing reliance on therapist supervision, and care services that hinder children from natural situations. However, there are many obstacles at present. In addition to insufficient resources, long waiting time for accessing services, and the COVID-19 Pandemic or future emerging infections interrupting in-person face-to-face services, remote guidance of parents to implement the intervention at home (telehealth) is another way to help children and families with developmental disabilities. This way of giving patients holistic health care is a new trend in providing early intervention services. Therefore, this study plans to first conduct team education and discussion, and then use our highly reliable screening tool to screen children aged 24-72 months for autism screening in the community and institutes. Those screened with a positive result will be referred to our early intervention center for comprehensive child development and behavioral follow-up. A total of 60 children over 24 months old diagnosed with ASD will participate in the telehealth intervention program. They will be randomly assigned to the intervention group or the comparison group. The intervention group (the telehealth group) will also receive a 16-week telehealth intervention with guidance, digital learning platform, teaching parents to learn intervention skills to improve children's attention and play ability, social communication, cognition, perceptual movement, and improve parents' management of children's behavior problems. The comparison group (telephone group) will receive 16-weeks of child development counseling through phone calls. This project aims to enhance the education and cooperation of the team, increase the awareness and understanding of ASD in the community, strengthen the use of relevant screening tools, provide an easy-accessed E-learning platform for parents, daycare or kindergarten caregivers or professionals to learn, and establish an evidence-based telehealth early intervention for autistic children. In this way, parents of autistic children would have more confidence and support to go for screening and intervention to achieve patient- and family-centered holistic care and enhance their compliance.

ELIGIBILITY:
Inclusion Criteria:

* child's age within 24-72 months
* parental age greater than 18 years
* parents have a minimum 9 years of education year that can read Chinese.

Exclusion Criteria:

* Children with major sensory, motor or neurological impairment/disorder (e.g., uncorrected visual or hearing loss, or severe brain damage)

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2024-08-18 (Estimated); Study Completion 2024-08-18 (Estimated)

PRIMARY OUTCOMES:
Mullen Scale of Early Learning (MSEL) | 16 weeks
  The MSEL assesses the child's developmental skills that provides standardized scores in five domains: Visual Reception, Receptive Language, Expressive Language, Fine Motor skills, and Gross Motor skills. The MSEL scores will be processed to examine the changes between the baseline and the post training.
Peabody Developmental Motor Scales, Second Edition (PDMS2) | 16 weeks
  The PDMS-2 is a norm-referenced assessment comprising 6 subscales, namely Reflexes, Locomotion, Object. The PDMS-2 scores will be processed to examine the changes between the baseline and the post training.
  Manipulation, Stationary, Grasping, and Visual-Motor Integration
Child Behavior Checklist for Ages 1.5-5 (CBCL/1.5-5) | 16 weeks
  The CBCL/1.5-5, a parental report of child behavioral, emotional and social functioning at ages 1.5-5 years, consists of 100 items. The CBCL/1.5-5 scores will be processed to examine the changes between the baseline and the post training.

SECONDARY OUTCOMES:
Parenting Stress Index (PSI) | 16 weeks
  The PSI is a 120-item, 5-point parent-report measure assessing parenting stress factors. The PSI scores will be processed to examine the changes between the baseline and the post training.
Satisfaction Questionnaire | 16 weeks
  Participating parents will be asked to complete a questionnaire assessing their satisfaction with the training that is specifically created for the purpose of the proposed study. The satisfaction questionnaire will only be filled out by participating parents at the time when complete all intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School and Graduate Institute of Physical Therapy, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No